CLINICAL TRIAL: NCT00874601
Title: Prospective, Randomized, Open-label, Blinded Endpoints, Multi-center Study to Evaluate the Efficacy of Modest Blood Pressure Reduction With Diovan® (Valsartan) in Acute Ischemic Stroke
Brief Title: Valsartan Efficacy on Modest Blood Pressure Reduction in Acute Ischemic Stroke
Acronym: VENTURE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VENTURE
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; blood pressure; valsartan; death; dependancy
MeSH Terms: conditions — Ischemic Stroke; Death | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- valsartan group (Experimental): The valsartan group will be initially given 80 mg of Diovan® (valsartan) per oral once daily in the morning on day 1, and flexibly will be adjusted to a dose of 80 -320 mg per day during next 6 days if more than 30% of SBPs measured at least 4 times in a day will not get the target level of SBPs.
  Interventions: Drug: Diovan® (valsartan)
- control group (No Intervention): Patients on control group will not receive any other antihypertensive medication for first 7 days after stroke onset. However, rescue therapy with antihypertensive agents can be permitted for episodes with severely elevated blood pressures during acute periods.

INTERVENTIONS:
Drug: Diovan® (valsartan) — The valsartan will be initially given 80 mg of Diovan® (valsartan) per oral once daily in the morning on day 1, and flexibly will be adjusted to a dose of 80 -320 mg per day during next 6 days if more than 30% of SBPs measured at least 4 times in a day will not get the target level of SBPs.
  In those patients not achieving target level of blood pressure (more than 15% reduction of initial blood pressure or below 145 mmHg of systolic blood pressure), an additional antihypertensive drugs (diuretics, beta blockers) can be given despite of Valsartan 320 mg. If the BP is considered to be low enough, dose of valsartan can be decreased to 40 mg per day. If the administration of valsartan is judged to be inappropriate by duty doctor due to any reasons, it can be stopped and the reasons will be recorded.
  Arms: valsartan group

SUMMARY:
The manipulation of blood pressure in acute cerebral ischemia has been a matter of debate until now. The investigators are clearly in need of more detailed data on how antihypertensive treatment affects outcome in acute phase of stroke.

This study will assess the effects of modest blood pressure (BP) lowering manipulation in acute period of ischemic stroke on death or dependency at 90-day.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients admitted within 24 hours and can be enrolled within 48 hours after qualifying ischemic stroke onset
* Patients with systolic blood pressure above 150 mm Hg and no more than 185 mm Hg at least twice of 3 or more times at 5 minutes intervals after resting
* Baseline NIHSS score at least 2 points, not more than 21 points
* Full functional independence prior to the present stroke indicated by an estimated premorbid mRS score of 0 or 1
* Informed consent from the patients or authorized representatives must be obtained in writing enrollment into the study

Exclusion Criteria:

* Patients who received thrombolytic therapy (intravenous or intraarterial)
* Patients with acute Intracerebral hemorrhage diagnosed by neuroimaging
* Patients with moderate or severe cardiac failure (New York Heart Association class III and IV)
* Patients with medical condition which need urgent or special antihypertentive therapy, such as hypertensive encephalopathy, aortic dissection, acute renal failure, acute pulmonary edema, or acute myocardial infarction
* Comatose at screening
* Known or suspected cerebral aneurysm or arteriovenous malformation
* Any other clinical relevant serious disease, including uncontrolled Diabetes, severe liver disease, or severe renal disease at the time of randomization
* Life expectancy of less than 3 months due to comorbid conditions, such as malignancy
* Participation in another drug trials or planned use of vascular interventions within the previous 30 days
* Women who are pregnant, breast feeding, or of child bearing potentials
* Contraindication to ARBs, such as history of angioedema to ARBs, renovascular hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Death or dependency measured as functional status with the use of mRDs | 90 days after the onset

SECONDARY OUTCOMES:
NIHSS | 7 days and 90 days after stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Byung-chul Lee, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Park TH, Lee JS, Park SS, Ko Y, Lee SJ, Lee KB, Lee J, Kang K, Park JM, Choi JC, Kim DE, Cho YJ, Kim JT, Kim DH, Cha JK, Han MK, Lee J, Oh MS, Yu KH, Lee BC, Bae HJ, Hong KS. Safety and efficacy of intravenous recombinant tissue plasminogen activator administered in the 3- to 4.5-hour window in Korea. J Stroke Cerebrovasc Dis. 2014 Aug;23(7):1805-12. doi: 10.1016/j.jstrokecerebrovasdis.2014.04.027. Epub 2014 Jun 21. PMID 24957314